CLINICAL TRIAL: NCT02735408
Title: Tensiomyography Effects of the Kinesiotape Tension in the Muscular Stiffness of the Low Back Region
Brief Title: Kinesiotape Tensiomyography in Low Back Region
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Monica Garcia, MSc,PT, Universidad Europea de Madrid
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P2015/35RM
Record Dates: First submitted 2015-12-18; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Bandages; Muscle Tonus; Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 100% KT Tension (Experimental): 100% KT Tension
  Interventions: Other: Kinesiotape (KT)
- 50% KT Tension (Experimental): 50% KT Tension
  Interventions: Other: Kinesiotape (KT)
- 0% KT Tension (Experimental): 0% KT Tension
  Interventions: Other: Kinesiotape (KT)
- Control (Without KT) (No Intervention): Control (Without KT)

INTERVENTIONS:
Other: Kinesiotape (KT)
  Arms: 0% KT Tension; 100% KT Tension; 50% KT Tension

SUMMARY:
Lumbar pain is a quite prevalent pathology in general population within general and sporting population, which comes to mean high sanitary and sport costs. This concrete pain´s nature is often unspecific, but it seems that one of the main risk factors that predispose to suffer from it are changes in the paravertebral-lumbar musculature stiffness.

Since one decade approximately, it has proliferated, especially within sportsmen and women the use of a therapeutic technique: the neuromuscular bandage best known as Kinesiotape (KT). This treatment seems to accept different applications, despite there´s still a lack of scientific evidence for several of its supposed effects. One of the theories about its use technique is that the bandage strain generates different effects in musculature stiffness. Thus, when the bandage is applied over the skin with a pre-stretching of the elastic bandage, it can cause arise of stiffness and strength muscle empowerment. On the other hand, if the bandage is applied without strain, the opposite result would appear, relaxation and strength muscle decrease.

For trainers and therapists is important to know if the KT effect differs over the bandage technique, since the application could be different according to the specific troubles reported by the athletes. For example, talking about cyclists, who keep constantly a hold rachis lumbar flexion, could be interesting to normalize the lumbar musculature stiffness, by placing the bandage with certain strain to achieve a mechanic effect. Nevertheless, talking about other sports like weightlifting, the bandage effect should be the stiffness arisen as a preventive measure, for avoiding injuries derived from the lack of motor control in the lumbar region. These lumbar-region muscle problems affect to popular and majority sports like football, so lumbar pain is very frequently reported by football players, normally due to an agonist-antagonist musculature unbalance. In all these terms, the use of KT would be interesting in order to reduce the musculature strain degree.

Tensiomyography (TMG) is showing as one of the most useful and reliable instrument for the musculature stiffness assessing, due to its velocity, harmlessness, sensing and high reproducibility. Taking in consideration that the maximum deformity measured by the TMG is inversely related with the muscle stiffness, and whereas this project pretends to modify that stiffness by means of the KT application, it seems obvious that TMG is the most suitable measurement instrument.

All these precedents considered, the present project pretends to analyze the effects of different KT strain application along 48 hours with strains techniques of 100%, strain 50% and strain 0% in the normalization of the paravertebral-lumbar musculature stiffness, by means of TMG monitoring.

DETAILED DESCRIPTION:
Lumbar pain is a quite prevalent pathology in general population within general and sporting population, which comes to mean high sanitary and sport costs. This concrete pain´s nature is often unspecific, but it seems that one of the main risk factors that predispose to suffer from it are changes in the paravertebral-lumbar musculature stiffness.

Since one decade approximately, it has proliferated, especially within sportsmen and women the use of a therapeutic technique: the neuromuscular bandage best known as Kinesiotape (KT). This treatment seems to accept different applications, despite there´s still a lack of scientific evidence for several of its supposed effects. One of the theories about its use technique is that the bandage strain generates different effects in musculature stiffness. Thus, when the bandage is applied over the skin with a pre-stretching of the elastic bandage, it can cause arise of stiffness and strength muscle empowerment. On the other hand, if the bandage is applied without strain, the opposite result would appear, relaxation and strength muscle decrease.

For trainers and therapists is important to know if the KT effect differs over the bandage technique, since the application could be different according to the specific troubles reported by the athletes. For example, talking about cyclists, who keep constantly a hold rachis lumbar flexion, could be interesting to normalize the lumbar musculature stiffness, by placing the bandage with certain strain to achieve a mechanic effect. Nevertheless, talking about other sports like weightlifting, the bandage effect should be the stiffness arisen as a preventive measure, for avoiding injuries derived from the lack of motor control in the lumbar region. These lumbar-region muscle problems affect to popular and majority sports like football, so lumbar pain is very frequently reported by football players, normally due to an agonist-antagonist musculature unbalance. In all these terms, the use of KT would be interesting in order to reduce the musculature strain degree.

Tensiomyography (TMG) is showing as one of the most useful and reliable instrument for the musculature stiffness assessing, due to its velocity, harmlessness, sensing and high reproducibility. Taking in consideration that the maximum deformity measured by the TMG is inversely related with the muscle stiffness, and whereas this project pretends to modify that stiffness by means of the KT application, it seems obvious that TMG is the most suitable measurement instrument.

All these precedents considered, the present project pretends to analyze the effects of different KT strain application along 48 hours with strains techniques of 100%, strain 50% and strain 0% in the normalization of the paravertebral-lumbar musculature stiffness, by means of TMG monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Subjets without exclusion criteria
* Workers from UEM

Exclusion Criteria:

* Low back conditions

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Tensiomyography changes (seconds): Delay time (Td) ; Contraction time (Tc) ; Sustain time (Ts) ; Relaxation time (Tr) | 4 Weeks
  Delay time (Td) as a time between the electrical impulse and 10% of the contraction; Contraction time (Tc) as a time between 10% and 90% of the contraction; Sustain time (Ts) as a time between 50% of the contraction and 50% of the relaxation; Relaxation time (Tr) as a time between 90% and 50% of the relaxation.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea, Madrid, Madrid, Spain